CLINICAL TRIAL: NCT02618785
Title: The Effect of Premedication Hyoscine-N-butylbromide Before Hysterosalpingography for Diagnosis of Proximal Tubal Obstruction in Infertile Women : A Randomized Double-Blind Controlled Trial
Brief Title: Antispasmodic Drug for Diagnosis Proximal Tubal Occlusion on Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Akarawit Jitchanwichai, Obstertrics and Gynecology department, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 562441242
Record Dates: First submitted 2015-11-21; First posted 2015-12-01 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2016-11

CONDITIONS: Tubal Obstruction
Keywords: Hysterosalpingography; antispasmodic drug; infertile women
MeSH Terms: conditions — Fallopian Tube Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyoscine (Experimental): The experiment group receive Hyoscine 10 mg 2 tablets by mouth before hysterosalpingography procedure
  Interventions: Procedure: hysterosalpingography
- Placebo (Placebo Comparator): The control group receive placebo by mouth before hysterosalpingography procedure
  Interventions: Procedure: hysterosalpingography

INTERVENTIONS:
Procedure: hysterosalpingography — Starting procedure by using largest appropriate speculum for maximum cervical exposure. Cleanse the cervix with povidone iodine. A tenaculum was applied to the anterior cervix to help for stabilization and counter-traction. Then insert a sterile Rubin's cannula into the cervix uteri. A scout radiograph of the pelvis was obtained with the catheter in place before contrast material was instilled. After that the water soluble contrast media was slowly instilled through the cannula appropriate volume range 10-15 ml., with fluoroscopic images obtained intermittently to evaluate the uterus, fallopian tubes and tubal patency
  Other Names: HSG

SUMMARY:
This study finds premedication Hyoscine-N-butylbromide before hysterosalpingography have a potential effect for diagnosis of proximal tubal obstruction in infertile women. The investigators did a double-blind, randomized placebo-controlled trial

DETAILED DESCRIPTION:
Infertility is a common gynecologic problem in reproductive medicine. The causes of female infertile can divided into ovulatory dysfunction, tubal and pelvic pathology, unexplained infertility and unusual problems. About 30-35% of case of infertility are caused by the tubal factor and tubal disease is an important cause of infertility and should be specifically excluded(1). Methods for evaluation of the fallopian tube pathology include the Hysterosalpingography(HSG), Saline infusion sonography(SIS) and Laparoscopy with chromopertubation etc(2-3).

Laparoscopy with chromopertubation is considered the definitive test for evaluating tubal disease and allows for the detection of other intraabdominal causes of infertility. However, laparoscopy is expensive, time consuming, limited in some centers, and unpleasant for the patient. More importantly many patients have anesthetic and surgical complications that require hospital admission(4). Therefore, HSG has been most commonly used for routine screening in infertility for evaluation of tubal patency. It is a simple, noninvasive and inexpensive technique. HSG is the standard first-line test to evaluate tubal patency(5-7).

HSG is an X-ray procedure that is used to view the inside of the uterus and fallopian tubes. HSG for investigating tubal patency has moderate sensitivity 65% but excellent specificity 83% in the infertile population. The PPV and NPV of HSG are 38% and 94%, respectively(8-9). However, it can have a false positive diagnosis if the HSG indicates occlusion, there may be a good chance 60% that the tubes are actually patent, and if the HSG demonstrates patency there is a little chance 5% that the tubes are occluded(10). There are several factors leading to a false diagnosis of tubal occlusion by using HSG. The most common factor cited is a cornual spasm(11), there could simply be a resistance difference between the two tubes(12) and the other factor are an existing of mucous plug at proximal part of the fallopian tube(13).

Diagnostic laparoscope performed after HSG showed a decrease in the rate of diagnoses of initial tubal occlusion by 40-60%(14-16). There are studies about repeat HSG 1 month later in patients whom HSG showed proximal tubal blockage, showed tubal patency about 60%(17). And there are many studies about administration of an antispasmodic or analgesic drug to distinguish tubal spasm from tubal occlusion during HSG. Such as Glucagon, Hyoscine butylbromide, ASA, Terbutaline, Diazepam, Fenoterol and Mitamizole etc(18-21). There is only one prospective study about hyoscine butylbromide use after tubal occlusion occur during HSG, showed that appears to be safe and effective drug to relieve proximal tubal obstruction by 80%(22).

Hyoscine-N-butylbromide(Buscopan®), an antispasmodic drug commonly used for relief of smooth muscle spasms and can use to relieve genito-urinary spasm. Hyoscine exerts a spasmolytic action, peripheral anticholinergic effects result from a ganglion-blocking action within the visceral wall as well as from anti-muscarinic activity, could decrease pain during uterine cramping. And about relief tubal obstruction in HSG procedure, no previous studies investigate compared its efficacy in randomized double-blind controlled trial. And there are inexpensive, safe with minimal side effects, then there are studies reported hyoscine can relieve dysmenorrhea too(23-24).

In Thailand, reported that one of the most common causes of female infertility is tubal pathology which accounted for 27% of the cases(25). And at Infertile clinic of Songklanagarind Hospital, mostly use HSG for standard first-line to evaluate tubal patency. We hypothesized that Hyoscine-N-butylbromide use before HSG can relieve the tubal occlusion that not true occlusion. It is possible to decrease the false positive rate of diagnosis of tubal occlusion cause from cornual spasm. So it can apply to use to decrease the necessity of laparoscopy with chromopertubation for definitive test tubal occlusion or repeated. And it will also reduce the medical cost of further more expensive investigation and medical complication.

ELIGIBILITY:
Inclusion Criteria:

* The infertile women who indicated for investigation hysterosalpingography were enrolled.

Exclusion Criteria:

1. Known sensitivity to Hyoscine or contrast media
2. Genital tract infection
3. Suspected pregnancy
4. Abnormal uterine bleeding

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
number result diagnosis of proximal tubal occlusion | up to 24 weeks
  To evaluate rate diagnosis of proximal tubal occlusion compare between Hyoscine group and placebo group before HSG.

SECONDARY OUTCOMES:
number of true occlusion or false occlusion | up to 24 weeks
  To evaluate false positive results of proximal tubal occlusion from HSG compare between study and control groups.
number of participants with treatment-related adverse effects of drug and procedure | up to 24 weeks
  such as dizziness, syncope, tachycardia, nausea, vomiting, pelvic pain, bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Akarawit Jitchanwicahi, MD, Study Director — Department of Obstetrics and Gynecology, Faculty of Medicine, Prince of Songkla University, Songkhla 90112, Thailand
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hindocha A, Beere L, O'Flynn H, Watson A, Ahmad G. Pain relief in hysterosalpingography. Cochrane Database Syst Rev. 2015 Sep 20;2015(9):CD006106. doi: 10.1002/14651858.CD006106.pub3. PMID 26387564
- [Background] Practice Committee of the American Society for Reproductive Medicine. Diagnostic evaluation of the infertile female: a committee opinion. Fertil Steril. 2015 Jun;103(6):e44-50. doi: 10.1016/j.fertnstert.2015.03.019. Epub 2015 Apr 30. PMID 25936238
- [Background] Steinkeler JA, Woodfield CA, Lazarus E, Hillstrom MM. Female infertility: a systematic approach to radiologic imaging and diagnosis. Radiographics. 2009 Sep-Oct;29(5):1353-70. doi: 10.1148/rg.295095047. PMID 19755600
- [Background] Hajishafiha M, Zobairi T, Zanjani VR, Ghasemi-Rad M, Yekta Z, Mladkova N. Diagnostic value of sonohysterography in the determination of fallopian tube patency as an initial step of routine infertility assessment. J Ultrasound Med. 2009 Dec;28(12):1671-7. doi: 10.7863/jum.2009.28.12.1671. PMID 19933481
- [Background] Kodaman PH, Arici A, Seli E. Evidence-based diagnosis and management of tubal factor infertility. Curr Opin Obstet Gynecol. 2004 Jun;16(3):221-9. doi: 10.1097/00001703-200406000-00004. PMID 15129051
- [Background] Moore DE. Pain associated with hysterosalpingography: Ethiodol versus Salpix media. Fertil Steril. 1982 Nov;38(5):629-31. doi: 10.1016/s0015-0282(16)46647-1. No abstract available. PMID 6290276
- [Background] Marjoribanks J, Ayeleke RO, Farquhar C, Proctor M. Nonsteroidal anti-inflammatory drugs for dysmenorrhoea. Cochrane Database Syst Rev. 2015 Jul 30;2015(7):CD001751. doi: 10.1002/14651858.CD001751.pub3. PMID 26224322
- [Background] Kemp JH. "Buscopan" in spasmodic dysmenorrhoea. Curr Med Res Opin. 1972;1(1):19-25. doi: 10.1185/03007997209111141. No abstract available. PMID 4589399
- [Background] Rohwer AC, Khondowe O, Young T. Antispasmodics for labour. Cochrane Database Syst Rev. 2013 Jun 5;2013(6):CD009243. doi: 10.1002/14651858.CD009243.pub3. PMID 23737030
- [Background] Alper MM, Garner PR, Spence JE. Hyoscine butylbromide to relieve utero-tubal obstruction at hysterosalpingography. Br J Radiol. 1985 Sep;58(693):915. doi: 10.1259/0007-1285-58-693-915-a. No abstract available. PMID 3842296
- [Background] Moro F, Selvaggi L, Sagnella F, Morciano A, Martinez D, Gangale MF, Ciardulli A, Palla C, Uras ML, De Feo E, Boccia S, Tropea A, Lanzone A, Apa R. Could antispasmodic drug reduce pain during hysterosalpingo-contrast sonography (HyCoSy) in infertile patients? A randomized double-blind clinical trial. Ultrasound Obstet Gynecol. 2012 Mar;39(3):260-5. doi: 10.1002/uog.11089. PMID 22223598
- [Background] Jareethum R, Suksompong S, Petyim S, Prechapanich J, Laokirkkiat P, Choavaratana R. Efficacy of mefenamic acid and hyoscine for pain relief during saline infusion sonohysterography in infertile women: a double blind randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2011 Apr;155(2):193-8. doi: 10.1016/j.ejogrb.2010.11.021. Epub 2010 Dec 30. PMID 21194827
- [Derived] Jitchanwichai A, Soonthornpun K. Effect of Premedication Hyoscine-N-Butylbromide before Hysterosalpingography for Diagnosis of Proximal Tubal Obstruction in Infertile Women: A Randomized Double-Blind Controlled Trial. J Minim Invasive Gynecol. 2019 Jan;26(1):110-116. doi: 10.1016/j.jmig.2018.03.034. Epub 2018 Apr 24. PMID 29702271